CLINICAL TRIAL: NCT04881162
Title: Feasibility Study of the Treatment of Acute Ischemic Stroke Using the NOVIS Transcarotid Neuroprotection System In Transcarotid Embolectomy
Brief Title: Feasibility Study of the Treatment of Acute Ischemic Stroke Using the NOVIS Transcarotid Neuroprotection System
Acronym: NITE1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to terminate study early solely due to slow enrollment.
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRM-2019-01
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
Keywords: mechanical thrombectomy; stroke treatment; embolic protection; transcarotid
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Patients with acute ischemic anterior circulation stroke due to large vessel embolic occlusion who are candidates for endovascular therapy and in whom transfemoral therapy failed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NOVIS Transcarotid Neuroprotection System (NPS) (Experimental): Patients that have failed transfemoral endovascular therapy in the case of anterior circulation strokes due to large vessel embolic occlusions will enrolled in the study and treated using the NOVIS Transcarotid NPS.
  Interventions: Device: NOVIS Transcarotid Neuroprotection System (NPS)

INTERVENTIONS:
Device: NOVIS Transcarotid Neuroprotection System (NPS) — The NOVIS Transcarotid Neuroprotection System (NPS) is intended to provide transcarotid vascular access and embolic protection

SUMMARY:
Study Objective is to establish the feasibility and safety of the NOVIS Transcarotid Neuroprotection System when used for the transcarotid intervention of patients that have a failed transfemoral endovascular therapy in the case of anterior circulation strokes due to large vessel embolic occlusions.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm feasibility study for the endovascular treatment of patients with acute ischemic anterior circulation strokes due to large vessel embolic occlusions using the transcarotid approach with flow reversal. Patients enrolled into the NITE 1 Study will have failed transfemoral therapy and will be followed immediately from post-op to 90 days.

ELIGIBILITY:
Inclusion Criteria Summary:

* 1. Patients presenting with acute ischemic stroke of the anterior circulation with large vessel occlusions who are eligible for revascularization using endovascular therapies (stentrievers and/or aspiration devices)

  2. Occlusion of the intracranial ICA, MCA M1, proximal MCA M2, single-vessel MCA M2, dominant MCA M2, or co-dominant MCA M2 segments

  3. Patient has failed transfemoral therapy (see Appendix 4 for definition), and at least 15 minutes have elapsed from groin puncture

Exclusion Criteria Summary:

* 1. Significant disease of the ipsilateral common carotid artery on routine CTA

  2. Presence of a cervical ICA loop or other high-risk anatomical features of the ICA on routine CTA, that may preclude the use of the NOVIS NPS

  3. Any active or recent hemorrhage within the past 30 days

  4. Embolectomy contraindications

  a. Pre-stroke mRS ≥2 b. NIHSS ≤ 5 c. ASPECTS ≤ 5

  5. IV tPA has been or is being administered

  6. Last known well > 24 hours ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Matouk, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Device-related Serious Adverse Events
Description: The primary outcome measure assesses the number of vascular complications which include which include dissection, pseudoaneurysm, hematoma, arteriovenous fistula, thrombus formation, embolization and any vascular complication that may be attributed to the device AND requires surgical repair, surgical wound revision, transfusion, etc. The endpoint is measured at 90 days post-procedure.
Time Frame: 90 Days
Measure: Number; unit: device-related serious adverse events
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
device-related serious adverse events | 0

2. Primary Outcome: Number of Other Serious Adverse Events
Description: The primary outcome measure assesses the number of permanent cranial nerve injury, new symptomatic ipsilateral hemorrhage and dissections related to ancillary devices. The endpoint is measured at 90 days post-procedure.
Time Frame: 90 Days
Measure: Number; unit: other serious adverse events
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
other serious adverse events | 0

3. Primary Outcome: Number of Subjects With Functional Independence
Description: Functional independence will be evaluated by assessing the modified Rankin scale (mRS). The mRS comprises six levels from 0 to 5 of increasing severe disability with an additional level 6 indicating death. A lower score indicates a better outcome and a higher score indicates a worse outcome. A mRS score reported between 0 to 2 will be considered functionally independent and 3 to 6 to not be functionally independent or dead at point of measurement. The endpoint is measured at 90 days post-procedure.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
Participants
  mRS of 0 to 2 | 4
  mRS of 3 to 6 | 8

4. Secondary Outcome: Carotid Access Time
Description: The endpoint measures the hospital arrival to neck incision, neck incision to carotid exposure, neck incision to carotid exposure, neck incision to carotid artery catheterization which includes the securement of the sheath, neck incision to femoral venous sheath access which includes the securement of the sheath, and neck incision to initiation of reverse flow.
Time Frame: Hospital arrival to neck incision, neck incision to carotid exposure, neck incision to carotid exposure, neck incision to carotid artery catheterization, neck incision to femoral venous sheath access which, and neck incision to initiation of reverse flow.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
minutes
  Hospital arrival to neck incision | 100.3 (40.6)
  Neck incision to carotid exposure | 13.5 (5.0)
  Neck incision to carotid catheterization (includes securement of sheath) | 20.4 (7.5)
  Neck incision to femoral venous sheath access (includes securement of sheath) | 6.8 (11.9)
  Neck incision to initiation of reverse flow | 35 (13.2)

5. Secondary Outcome: Time to Final Revascularization
Description: The endpoint measures the time of hospital arrival to operating room (OR), last known well to final revascularization, admission to final revascularization, OR to final revascularization, Cutdown to final revascularization, arterial introduction of interventional tools to final revascularization, total reverse flow time including common carotid artery (CCA) clamp to CCA unclamp.
Time Frame: Hospital arrival to OR, LKW to final revascularization, admission to final revascularization, OR to final revascularization, cutdown to final revascularization, arterial introduction of interventional tools to final revascularization, total reverse flow.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
minutes
  Hospital arrival to operating room | 46.7 (41.9)
  Last known well to final reperfusion | 628.9 (336.0)
  Admission to final reperfusion | 156.7 (32.0)
  Operating room to final reperfusion | 110.0 (43.05)
  Cutdown to final reperfusion | 56.3 (25.1)
  Arterial introduction of interventional tools to final reperfusion | 22.0 (24.2)
  Total reverse flow time (CCA clamp to CCA unclamp) | 20.3 (26.2)

6. Secondary Outcome: Number of Device-Related Complications
Description: This outcome measure assesses the number of reported complications that may be attributed to the device through the end of all patient follow up in the study.
Time Frame: 90 Days
Measure: Number; unit: complications
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
complications | 1

7. Secondary Outcome: Neurologic Assessment
Description: The outcome measure measures neurological worsening of patients according to the National Institutes of Health Stroke Scale (NIHSS) at 90 days post procedure. The NIHSS is a graded neurological examination that assesses consciousness, eye movements, visual fields, motor and sensory impairments, ataxia, speech, cognition and inattention. The NIHSS is a combination of 11 components each with a particular scale as follows: level of consciousness (1a: 0-3, 1b: 0-2 and 1c: 0-2), best gaze (0-2), visual fields (0-3), facial palsy (0-3), arm motor (0-4), leg motor (0-4), limb ataxia (0-2), sensory (0-2), best language (0-3), dysarthria (0-2), extinction and inattention (0-2). The components are summed, and a lower score indicates better outcomes, and higher score indicates worse outcomes. A neurological worsening similar to a non-disabling stroke is considered scored less than or equal to 4 and a neurological worsening similar to a disabling stroke with a score equal to or greater than 5.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
Participants
  Non-Disabling Stroke (NIHSS ≤ 4) | 8
  Disabling Stroke (NIHSS ≥ 5 | 4

8. Secondary Outcome: Technical Sucess Rate
Description: The outcome measure will count the number patients with successful introduction of endovascular tools through the NOVIS Transcarotid NPS during the procedure. Introduction of endovascular tools will be considered successful if NPS was placed, reverse flow was established, and interventional tools were successfully delivered.
Time Frame: Start to end of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
Participants
  Technical Sucess Achieved | 12
  Technical Sucess Not Achieved | 0

9. Secondary Outcome: Revascularization Sucess Rate
Description: The outcome measure reports the number of patients with modified thrombolysis in cerebral infarction (mTICI) score evaluated by the contract core lab measuring angiograms collected from baseline to immediately after the end of the index procedure. The mTICI grading scale is a tool for determining the response of thrombolytic therapy for ischemic stroke on a scale between 0 to 3. A lower score indicates better outcomes and higher score indicates worse outcomes The score 2 has two additional grades of severity of 2a and 2b indicating worse outcomes along the alphabetical progression of the scale.
Time Frame: Start to end of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
Number analyzed (Participants) | 12
Participants
  mTICI score 2b | 10
  mTICI score 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 90 days follow up post procedure
Description: Subjects who underwent the NOVIS Transcarotid NPS are included in the analysis set. Subjects who did not undergo the NOVIS Transcarotid NPS are excluded from analysis.
Arm/Group | NOVIS Transcarotid Neuroprotection System (NPS)
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOVIS Transcarotid Neuroprotection System (NPS) (N=12)
Death (General disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Reperfusion injury (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOVIS Transcarotid Neuroprotection System (NPS) (N=12)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Delirium (Psychiatric disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Asthenia (General disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Cytotoxic edema (Nervous system disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Genital injury (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Atrial enlargement (Cardiac disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Administration site hematoma (General disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Sponsor decided to terminate study early solely due to slow enrollment leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT04881162/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04881162/SAP_001.pdf